CLINICAL TRIAL: NCT01311115
Title: Using Group Commitment for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Srinakharinwirot University (Other)
Responsible Party: Principal Investigator, William Dow, Henry J. Kaiser Professor of Health Economics, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-04-1269; 2P30AG012839-16 (NIH); R21HD056581 (NIH)
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Results first posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group commitment contracts (Experimental): In addition to education and counseling, the intervention includes the following components:
  1. Each participant is encouraged to deposit his "cigarette money" on a weekly basis, to be returned only if the smoker quits successfully within three months.
  2. The project gives a series of two matching contributions of 150 baht each to participants who meet certain deposit requirements.
  3. Each participant is paired with another study participant. If both quit, each receives a cash bonus of 1,200 baht. At enrollment, pairs receive brief counseling on ways to support each other during the quit attempt.
  Interventions: Behavioral: Group commitment contract; Behavioral: Smoking cessation education and counseling
- Education and counseling (Active Comparator): Participants in this group receive educational pamphlets about quitting smoking and one-time, group counseling from a nurse trained in smoking cessation counseling.
  Interventions: Behavioral: Smoking cessation education and counseling

INTERVENTIONS:
Behavioral: Group commitment contract — 1. Each participant is required to deposit at least 50 baht at enrollment. A deposit collector visits each participant on a weekly basis and collects additional deposits on a voluntary basis. All deposits are returned only if the smoker quits successfully within three months.
  2. The project gives a matching contribution of 150 baht for the initial deposit of at least 50 baht. All participants in the treatment group are further randomized to a one-month group and a three-month group. The one-month group receives an additional 150 baht of project funds if they deposit 100 baht of their money within one month of enrollment. The three-month group receives 150 baht for depositing 100 baht within three months of enrollment.
  3. Each participant is paired with another study participant. If both quit, each receives a cash bonus of 1,200 baht. At enrollment, pairs receive brief counseling on ways to support each other during the quit attempt.
  Other Names: Commitment contract; Deposit contract; Contingency contract; Buddy intervention; Partner intervention
  Arms: Group commitment contracts
Behavioral: Smoking cessation education and counseling — Participants receive educational pamphlets on reasons to quit smoking and strategies for quitting smoking. They also receive one-time, group counseling on quitting smoking from a nurse trained in smoking cessation counseling.
  Other Names: Smoking cessation counseling

SUMMARY:
This study proposes a novel behavioral intervention to help smokers in Thailand to achieve their goals of quitting. Smoking treatment programs are rare throughout most of Asia and unlikely to meet the impending demand for quitting that tobacco control regulations is stimulating. New approaches are needed.

The present study is a randomized controlled trial to test the effectiveness of a novel, scalable approach to smoking cessation that is targeted toward rural Southeast Asian communities. Thailand is used as a test case to explore if pairs of smokers quit successfully after making financially-backed commitments and receiving cash incentives to quit. The control group receives education and counseling about quitting. In addition to education and counseling about quitting, the intervention includes two key components:

1. Each participant is encouraged to deposit his "cigarette money" on a weekly basis, to be returned only if the smoker quits successfully within three months. Such commitment contracts, based on theory from behavioral economics, are designed to help a person to maintain self-control and motivation in the face of temptation.
2. Each participant is paired with another study participant. If both quit, each receives a cash bonus. The joint incentives are designed to lead partners to support each other throughout the quit attempt.

Thus, group commitment contracts marshal a robust blend of elements: financial commitment, social support, peer pressure, and monetary rewards. A larger, follow-up evaluation will clarify the relative importance of each of these elements.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker of at least 10 cigarettes per week and at least 100 cigarettes over the course of a lifetime
* Residents of the study area in Nakhon Nayok province, which includes the six subdistricts of Klong Yai, Chumpon, Bueng San, Pak Phli, Khao Phoem, or Ongkharak

Exclusion Criteria:

* Pregnant
* Plans to leave the study area within the next 12 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin S White, MA, MSPH, Study Director — University of California at Berkeley; William H Dow, PhD, Principal Investigator — University of California at Berkeley; Suthat Rungruanghiranya, MD, Study Director — Srinakharinwirot University
Locations (1):
- Srinakharinwirot University, Ongkharak, Changwat Nakhon Nayok, Thailand

REFERENCES:
- [Result] White JS, Dow WH, Rungruanghiranya S. Commitment contracts and team incentives: a randomized controlled trial for smoking cessation in Thailand. Am J Prev Med. 2013 Nov;45(5):533-42. doi: 10.1016/j.amepre.2013.06.020. PMID 24139765

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Commitment Contracts: The intervention includes the following components:
  1. Education and counseling (same as control group): Participants receive educational pamphlets on reasons to quit smoking and strategies for quitting smoking. They also receive one-time, group counseling on quitting smoking from a nurse trained in smoking cessation counseling.
  2. Each participant is required to deposit at least 50 baht at enrollment. A deposit collector visits each participant on a weekly basis and collects additional deposits on a voluntary basis. All deposits are returned only if the smoker quits successfully within three months.
  3. The project gives a matching contribution of 150 baht for the initial deposit of at least 50 baht. All participants in the treatment group are further randomized to a one-month group and a three-month group. The one-month group receives an additional 150 baht of project funds if they deposit 100 baht of their money within one month of enrollment. The three-month group receives 150 baht for depositing 100 baht within three months of enrollment.
  4. Each participant is paired with another study participant at enrollment. If both quit, each receives a cash bonus of 1,200 baht. At enrollment, pairs receive brief counseling on ways to support each other during the quit attempt.
Period: Overall Study
Arm/Group | Group Commitment Contracts | Education and Counseling
Started | 132 | 69
Completed | 132 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Commitment Contracts | Education and Counseling | Total
Number analyzed (Participants) | 132 | 69 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.05 (13.82) | 51.07 (14.04) | 51.06 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 116 | 60 | 176
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Thailand | 132 | 69 | 201
Religion [Count of Participants; unit: Participants] — Population: Missing baseline data
  Participants
    number analyzed (Participants) | 131 | 69 | 200
    Buddhist | 91 | 48 | 139
    Muslim | 40 | 21 | 61
Education (years) [Count of Participants; unit: Participants] — Population: Missing baseline data
  Participants
    number analyzed (Participants) | 131 | 69 | 200
    0-3 years | 62 | 34 | 96
    4-6 years | 29 | 22 | 51
    7 or more years | 40 | 13 | 53
Monthly household income [Mean (Standard Deviation); unit: USD, in 100s] — Population: Missing baseline data
  USD, in 100s
    number analyzed (Participants) | 131 | 69 | 200
    (all) | 4.011 (5.805) | 3.513 (2.809) | 3.838 (4.971)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Status at 6 Months
Description: 7-day point prevalence of smoking abstinence measured 6 months after enrollment, using a NicCheck urine cotinine test. Participants who self-report having smoked in the last 7 days, as part of the follow-up survey, are considered to be continuing smokers.
Time Frame: 6 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group Commitment Contracts | Education and Counseling
Number analyzed (Participants) | 128 | 68
Participants | 57 | 13

2. Secondary Outcome: Concordance of Smoking Status Between Partners at 6 Months
Description: The concordance of smoking status among randomly assigned pairs: both abstain, both smoke, or one abstains and one smokes, measured using 7-day point-prevalence abstinence at 6 months after enrollment, measured using self-reported abstinence and urine cotinine testing. Participants in the control condition are assigned to a pair, but their partner's identity is never revealed during the study.
Time Frame: 6 months after enrollment
Population: In the education and counseling group, this represents a partner who is randomly assigned to the person but whose identity is never revealed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Commitment Contracts | Education and Counseling
Number analyzed (Participants) | 127 | 55
Participants
  Both abstain | 31 | 2
  Both smoke | 45 | 36
  One abstains, one smokes | 51 | 17

3. Secondary Outcome: Smoking Status at 3 Months
Description: 7-day point prevalence of smoking abstinence measured 3 months after enrollment, using a NicCheck urine cotinine test. Participants who self-report having smoked in the last 7 days, as part of the follow-up survey, are considered to be continuing smokers.
Time Frame: 3 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group Commitment Contracts | Education and Counseling
Number analyzed (Participants) | 128 | 68
Participants | 60 | 10

4. Secondary Outcome: Concordance of Smoking Status Between Partners at 3 Months
Description: The concordance of smoking status among randomly assigned pairs: both abstain, both smoke, or one abstains and one smokes, measured using 7-day point-prevalence abstinence at 3 months after enrollment, measured using self-reported abstinence and urine cotinine testing. Participants in the control condition are assigned to a pair, but their partner's identity is never revealed during the study.
Time Frame: 3 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group Commitment Contracts | Education and Counseling
Number analyzed (Participants) | 128 | 55
Participants
  Both abstain | 35 | 0
  Both smoke | 44 | 40
  One abstains, one smokes | 49 | 15

5. Secondary Outcome: Smoking Status at 14 Months
Description: as for outcome 1
Time Frame: 14 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group Commitment Contracts | Education and Counseling
Number analyzed (Participants) | 128 | 68
Participants | 53 | 17

ADVERSE EVENTS:
Arm/Group | Group Commitment Contracts | Education and Counseling
All-Cause Mortality (participants affected / at risk) | 1/132 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/69
Other Adverse Events (participants affected / at risk) | 0/132 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No